CLINICAL TRIAL: NCT06055595
Title: The Impact of Genetic Factors on Pregnancy Outcomes in Chronic Pancreatitis
Brief Title: Genetic Factors and CP Pregnancy Outcomes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CP-gene-pregnancy outcomes
Record Dates: First submitted 2023-09-13; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chronic Pancreatitis; Genetic Mutation; Pregnancy Related
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Years
Biospecimen Retention: Samples With DNA — The remained peripheral blood sample after laboratory examinations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: genetic sequencing — sequencing the susceptibility genes for CP, including serine protease inhibitor Kazal type 1, cationic trypsinogen, cystic fibrosis transmembrane conductance regulator, chymotrypsin C, etc.

SUMMARY:
To explore the impact of chronic pancreatitis (CP) susceptibility genes on pregnancy outcomes.

DETAILED DESCRIPTION:
The goal of this observational study is to explore the impact of CP susceptibility genes (SPINK1, PRSS1, CTRC, CFTR) on pregnancy outcomes (including both maternal and fetal outcomes) in a large Chinese cohort. Participants will be asked to provide their pregnancy-related data.

ELIGIBILITY:
Inclusion Criteria:

* female patients with a diagnosis of chronic pancreatitis
* have known genetic backgrounds and pregnancy history
* agree to join the study and provide informed consent

Exclusion Criteria:

* patients without documented pregnancy
* patients who denied to provide pregnancy-related information, or with incomplete pregnancy characteristics and/or outcomes
* patients with other autoimmune comorbidities that might influence pregnancy outcomes, such as systemic lupus erythematosus, autoimmune thyroid diseases, etc

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There were 292 female patients diagnosed with CP and underwent genetic testing from January 2010 to December 2014 in this cohort. After application of exclusion criteria, a total of 160 patients who had known genetic backgrounds and pregnancy history were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
adverse maternal outcomes of female CP patients | through study completion, an average of 1 year
  * CP-associated caesarean delivery referred to caesarean deliveries which happened due to the attack of CP or comorbidities associated with CP such as GDM and HDP.
  * CP-associated preterm delivery was defined as preterm deliveries which happened due to the attack of CP or comorbidities associated with CP.
  * GDM was defined as the onset or first recognition of abnormal glucose tolerance during pregnancy.
  * Intrahepatic cholestasis of pregnancy was based on characteristic symptoms, as well as elevated serum bile acids, in the absence of other hepatobiliary disease.
  * HDP included preeclampsia/eclampsia, chronic hypertension, chronic hypertension with superimposed preeclampsia, and gestational hypertension.
adverse fetal outcomes of female CP patients | through study completion, an average of 1 year
  * Low birth weight was defined as weight at birth <2500 g.
  * CP-associated abortion referred to abortions (i.e., a nonviable intrauterine pregnancy up to 20 weeks' gestation) which happened due to the attack of CP or comorbidities associated with CP.
  * Congenital anomaly referred to the inborn errors of development.
  * Stillbirth was defined as the delivery of a fetus ≥20 weeks of gestation with no signs of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wu D, Ru N, Wang YC, Ma GX, Shi TY, Xiong SH, You AJ, Wang L, Hu LH, Li ZS, Zou WB, Liao Z. Genetic Factors Associated With Adverse Pregnancy Outcomes in Chronic Pancreatitis. Clin Transl Gastroenterol. 2024 Apr 1;15(4):e00691. doi: 10.14309/ctg.0000000000000691. PMID 38334943